CLINICAL TRIAL: NCT05326867
Title: Comparison of Infiltration of 2% Lidocaine With and Without Needle as Analgesia in Epidural Needle Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Raden Besthadi Sukmono, Anesthesiologist, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IF
Record Dates: First submitted 2022-03-28; First posted 2022-04-14 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Epidural; Anesthesia, Headache; Analgesia
Keywords: Lidocaine infiltration; Epidural needle insertion; Epidural anesthesia.
MeSH Terms: conditions — Headache; Agnosia | interventions — Needles

STUDY DESIGN:
Intervention Model Description: This study was a double blind randomized controlled trial. Data collection was carried out consecutively on 84 subjects with 42 subjects in each group of lidocaine infiltration without needles and lidocaine infiltration with 23G needles
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, care providers, and investigators are blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Infiltration of 2% Lidocaine with Needle (Active Comparator): Free needle infiltration of lidocaine can be an alternative to reduce epidural needle insertion pain. The study of Gozdemir et al. found that 10% lidocaine infiltration without needle was less painful than 2% lidocaine infiltration with a 27G needle with no significant difference in analgesia effect during epidural needle insertion. This study aimed to compare infiltration of lidocaine with and without needle for epidural needle insertion
  Interventions: Device: Infiltration of 2% Lidocaine with Needle
- Infiltration of 2% Lidocaine without Needle (Active Comparator): Free needle infiltration of lidocaine can be an alternative to reduce epidural needle insertion pain. The study of Gozdemir et al. found that 10% lidocaine infiltration without needle was less painful than 2% lidocaine infiltration with a 27G needle with no significant difference in analgesia effect during epidural needle insertion. This study aimed to compare infiltration of lidocaine with and without needle for epidural needle insertion
  Interventions: Device: Infiltration of 2% Lidocaine without Needle

INTERVENTIONS:
Device: Infiltration of 2% Lidocaine with Needle — Infiltration of 2% Lidocaine with Needle
  Arms: Infiltration of 2% Lidocaine with Needle
Device: Infiltration of 2% Lidocaine without Needle — Free needle infiltration of lidocaine can be an alternative to reduce epidural needle insertion pain. The study of Gozdemir et al. found that 10% lidocaine infiltration without needle was less painful than 2% lidocaine infiltration with a 27G needle with no significant difference in analgesia effect during epidural needle insertion. This study aimed to compare infiltration of lidocaine with and without needle for epidural needle insertion
  Arms: Infiltration of 2% Lidocaine without Needle

SUMMARY:
One way to reduce pain during epidural needle insertion is infiltration of lidocaine using a needle. However, infiltration of lidocaine using the needle alone is a painful process. Free needle infiltration of lidocaine can be an alternative to reduce epidural needle insertion pain. The study of Gozdemir et al. found that 10% lidocaine infiltration without needle was less painful than 2% lidocaine infiltration with a 27G needle with no significant difference in analgesia effect during epidural needle insertion. This study aimed to compare infiltration of lidocaine with and without needle for epidural needle insertion in a double-blind study, using a Tuohy needle, Comfort-inTM injector, and wider surgical group as novelty from previous studies.

This study was a double blind randomized controlled trial. Data collection was carried out consecutively on 84 subjects with 42 subjects in each group of lidocaine infiltration without needles and lidocaine infiltration with 23G needles. The effectiveness of analgesia was assessed from three variables like pain with a Numeric Pain Rating Scale (NPRS) of 0 to 10 during lidocaine infiltration, pain with NPRS during epidural needle insertion, and patient movement during epidural needle insertion.

DETAILED DESCRIPTION:
Pain control is an important aspect in patient who will undergo a medical procedure. Reducing pain will not only improves patient satisfaction and comfort, but also provide speedy and easy medical procedures application. One of the patient's concerns regarding Anesthesia is pain when needles injected intracutaneously, intramuscularly, intravenously, or intrathecally. Epidural anesthesia is one of the neuraxial block technique resulting in sympathetic, sensory, and motor block depending on the dose, concentration, and volume of the local anesthetic administered. Epidural anesthesia was performed in 118 cases (18%) of the total 672 anesthesia cases in November 2020 at the National Central General Hospital (RSUPN) Cipto Mangunkusumo. Tuohy Type is one of epidural needles commonly used in Epidural anesthesia at Cipto Mangunkusumo General Hospital. This needle's size is large enough so that it causes pain if local anesthetic is not given prior to insertion. One of the way to administer local anesthetic prior to epidural needle insertion is by skin infiltration using a needle.

Ramzi in his research found that the median Visual Analogue Scale (VAS) due to epidural needle insertion given lidocaine infiltration with a needle is 5 with a range of 0-10. Mogensen investigated differences in pain expectations and the actual pain experienced by the patient due to insertion of the Tuohy needle in epidural anesthesia infiltrated with lidocaine using a needle. The research found that the median Numeric Rating Scale (NRS) for pain expectations was 5 while the NRS for actual pain experienced by patients was 2 (p value < 0.0001). Infiltration of local anesthetic with the needle alone is painful. Gozdemir in his research found that the pain median due to infiltration lidocaine using the needle before insertion of the epidural needle was 2 with a range of 0 up to 4.

Several alternative methods have been developed to reduce the pain of local anesthetic infiltration prior to epidural needle insertion, such as: establishing good communication with the patient during the procedure, replacing local anesthetic agents with chloroprocaine, adding bicarbonate to make lidocaine pH close to physiological pH, cooling down the skin with cryoanalgesia, local anesthetic infiltration with a smaller needle (25-30 G needle), lidocaine patch, and Eutectic Mixtures of Local Aesthetics (EMLA). Some of these alternatives still perform needle punctures that can produce pain, although to a lesser degree, and 10% of the population have a needle phobia. Non-invasive alternatives such as EMLA or cryoanalgesia cannot be a thorough solution due to the depth of analgesia generated. A study stated that the depth from skin to lumbar epidural cavity in parturient is 2-9 cm with 89% being on the 3.5-7.5 cm intervals. In leaner patients, the depth of the lumbar epidural found at 2-4 cm. Whereas EMLA only provides analgesia in depth of 2.9-4.5 mm if EMLA is applied for 60-120 minutes and 6 mm if applied for 3-4 hours. While cryoanalgesia such as vapocoolants spray works as a temporary topical analgesia by cooling the skin thereby reducing the sensitivity of pain receptors.

Needle usage, the length of time it takes to produce analgesia, transient analgesia results, and lack of depth of analgesia are the problems to present an alternative to local anesthetic infiltration that is completely pain free and adequate. A needleless injection technology can be a solution to these problems. The medicinal liquid is injected by a tool with high speed and pressure through a smooth hole. This system is expected to make the analgesia condition can be achieved quickly, painlessly, and avoiding needle phobia

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery patients undergoing epidural anesthesia (from thoracic 11 to lumbar 5) at Cipto Mangunkusumo General Hospital
* Patients aged 19 to 65 years
* Patients with American Society of Anaesthesiologist (ASA) criteria 1 to 3
* Willing to participate and signing the agreement

Exclusion Criteria:

* Epidural anesthesia with combined spinal epidural needle (Espocan)
* Epidural anesthesia is contraindicated
* Patients with a history of local anesthetic allergy
* The patient who cannot sit or feels pain when in a sitting position

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Pain Scale (NPRS scale) when Lidocaine Infiltrated | Immediately after Lidocaine is infiltrated
  The pain measurement with NPRS scale when 2% Lidocaine infiltrated
Pain Scale (NPRS scale) when Epidural Needle Inserted | Immediately after Epidural Needle Inserted
  The pain measurement with NPRS scale when Epidural Needle Inserted
Patient's Movement when Lidocaine Infiltrated | Immediately after Lidocaine is infiltrated
  Observation of patient's movement when 2% Lidocaine infiltrated
Patient's Movement when Epidural Needle Inserted | Immediately after Epidural Needle Inserted
  Observation of patient's movement when Epidural Needle Inserted

CONTACTS AND LOCATIONS:
Overall Officials: Raden B Sukmono, Principal Investigator — Indonesia University
Locations (1):
- RSUPN Cipto Mangunkusumo, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No